CLINICAL TRIAL: NCT03106571
Title: Phase 1 Safety-interaction Study of Pomaglumetad Methionil for Methamphetamine Use Disorder
Brief Title: Study of Pomaglumetad and Methamphetamine
Acronym: POMA-MA-Ph1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Deemed unable to enroll targeted participants in part due to COVID-19 shut downs
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Keith Heinzerling, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01DA043238 (NIH); R01DA043238 (NIH)
Record Dates: First submitted 2017-03-07; First posted 2017-04-10 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Methamphetamine Use Disorder
Keywords: Phase 1 clinical trial
MeSH Terms: interventions — pomaglumetad methionil; Methamphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pomaglumetad methionil Low + Methamphetamine (Experimental): Pomaglumetad 40 mg orally twice daily x 9 days with intravenous methamphetamine challenges
  Interventions: Drug: Pomaglumetad methionil; Drug: Methamphetamine
- Pomaglumetad methionil Mid + Methamphetamine (Experimental): Pomaglumetad 40 mg orally twice daily x 1 day then pomaglumetad 80 mg orally twice daily x 8 days with intravenous methamphetamine challenges
  Interventions: Drug: Pomaglumetad methionil; Drug: Methamphetamine
- Pomaglumetad methionil High + Methamphetamine (Experimental): Pomaglumetad 40 mg orally twice daily x 1 day then pomaglumetad 160 mg orally twice daily x 8 days with intravenous methamphetamine challenges
  Interventions: Drug: Pomaglumetad methionil; Drug: Methamphetamine
- Control + Methamphetamine (Placebo Comparator): 1-4 placebo tabs orally twice daily x 9 days (to match pomaglumetad dosing in each cohort) with intravenous methamphetamine challenges
  Interventions: Drug: Placebo; Drug: Methamphetamine

INTERVENTIONS:
Drug: Pomaglumetad methionil — Tablets twice daily
  Arms: Pomaglumetad methionil High + Methamphetamine; Pomaglumetad methionil Low + Methamphetamine; Pomaglumetad methionil Mid + Methamphetamine
Drug: Placebo — 1-4 tablets twice daily
  Arms: Control + Methamphetamine
Drug: Methamphetamine — intravenous methamphetamine

SUMMARY:
This is the first study of pomaglumetad in humans using methamphetamine. The goal of the study is to determine if pomaglumetad is safe when administered with methamphetamine. If shown to be safe with methamphetamine in the current study, a phase 2 clinical trial of pomaglumetad would be done to begin to find out if pomaglumetad is effective in treating methamphetamine use disorder.

DETAILED DESCRIPTION:
The study design is a randomized, double-blind, placebo-controlled multiple ascending-dose study of pomaglumetad in 24 non-treatment seeking participants with methamphetamine use disorder. Three cohorts of 8 participants each (total N = 24) will be enrolled and within each cohort participants will be randomly assigned in a 6:2 ratio to undergo methamphetamine infusions and assessments during treatment with pomaglumetad (N = 6 per cohort) or placebo (N = 2 per cohort). Participants in cohort 1 will receive pomaglumetad 40 mg orally twice daily (BID) or placebo, cohort 2 will receive pomaglumetad 80 mg BID or placebo, and cohort 3 will receive pomaglumetad 160 mg BID or placebo.

After completing outpatient baseline and screening/eligibility assessments, eligible participants will be admitted to the UCLA Hospital and will remain hospitalized during all experimental procedures (approximately 11 days and 10 nights).

A urine drug toxicology screen free of illicit substances (with the exception of THC) is required for admission. Upon admission, participants will receive a sample/test infusion of MA 30 mg IV. Participants tolerating the test infusion (no serious adverse advents and not exceeding stopping criteria below) will be randomized to receive POMA (40 mg BID in cohort 1, 80 mg BID in cohort 2, and 160 mg BID in cohort 3) or placebo.

Following three days of MA abstinence and POMA/placebo dosing to achieve study medication steady-state, participants will complete a MA self-administration session.

After two days for MA washout, participants will then have serial plasma samples collected over 12 hours to assess PK for POMA. The next day, participants will receive a 30 mg MA infusion followed by serial plasma sample collection over the following 48 hours for MA PK analysis.

Measures of cardiovascular response, subjective effects, and adverse events will be assessed following all MA infusions during self-administration and PK sessions.

Upon completion of the PK sample collection, participants will be discharged and a 14-day post-discharge (± 7 days) follow-up outpatient visit will be completed for safety purposes.

ELIGIBILITY:
Inclusion Criteria:

1. not seeking treatment for MA problems at the time of the study;
2. English-speaking;
3. age 18-55 years inclusive;
4. meet DSM-5 criteria for MA use disorder, moderate-severe as diagnosed via MINI;
5. have a self-reported history of using MA either via injection or smoking and provide at least one MA-positive urine prior to admission;
6. provide a urine drug screen negative for all illicit drugs, excepting THC, on the day of scheduled inpatient admission;
7. report methamphetamine use on 10 or more days in the past 30 days at baseline;
8. have a resting heart rate ≤ 100 bpm, systolic blood pressure ≤ 160 mm Hg, and diastolic blood pressure ≤ 100 mm Hg prior to admission;
9. have a baseline EKG that demonstrates normal sinus rhythm, QTc ≤ 450 msec in men or QTc ≤ 460 msec in women, and no clinically significant arrhythmias;
10. if female (except females of non-childbearing potential-e.g., at least 1 year post-menopausal or surgically sterile), not pregnant confirmed by negative pregnancy test nor lactating and willing to use a medically approved method of birth control to prevent pregnancy during the trial and for 40 days after the last dose of study medication;
11. if male, willing to refrain from donating sperm during the study and for 100 days following the last dose of study medication and agree that they and their partners will use a medically approved contraceptive method;
12. have a medical history and physical/neurological examination demonstrating no additional clinically significant contraindications for study participation, in the judgment of the investigators;
13. able to participate in all scheduled evaluations, likely to complete all scheduled tests, and likely to be adherent, in the opinion of the investigator and;
14. agree not to post any personal medical data or information related to the study on any social media site or website until the trial has completed.

Exclusion Criteria:

1. non-English speaking;
2. currently on probation or parole;
3. have current cocaine, opioid, marijuana, or alcohol use disorder, moderate-severe;
4. have liver function tests (total bilirubin, ALT, AST, or alkaline phosphatase) ≥ 2 x the upper limit of normal or kidney function tests (creatinine and BUN) ≥ 2 x the upper limit of normal;
5. current or past history of seizure disorder;
6. a history of head trauma that resulted in neurological sequelae;
7. major psychiatric disorder not due to substance abuse (e.g., schizophrenia, bipolar illness but excepting stable major depressive disorder, generalized anxiety disorder, etc.) as assessed by the MINI;
8. have a current neurological disorder (e.g., organic brain disease, dementia) or medical condition which would make study compliance difficult or compromise informed consent;
9. current ongoing treatment with psychotropic medications (e.g. antidepressants, antipsychotics, antiepileptics, sedative/hypnotics, narcotic analgesics);
10. history of suicide attempt(s) in the past 6 months or active suicidal intention or plan (score 4 or 5) in the past month as assessed by the C-SSRS;
11. evidence of clinically significant heart disease or hypertension;
12. evidence of untreated or unstable serious medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease including active tuberculosis infection;
13. have HIV infection and currently symptomatic, have a diagnosis of AIDS, or are receiving antiretroviral medication;
14. have a medical condition that makes maintaining reliable intravenous access impossible;
15. donated blood or plasma within 3 months of inpatient admission;
16. use of OAT1 inhibitor (e.g. probenecid, uricosurics, antivirals, nonsteroidal anti-inflammatories, loop diuretics, angiotensin II receptor antagonists, proton pump inhibitors, or statins) or CYP2D6 inducers or inhibitors within 14 days or five half-lives, whichever is longer, from admission;
17. currently employed by UCLA or Denovo or a first-degree relative of UCLA or Denovo employee or;
18. any other circumstances that, in the opinion of the investigators, would compromise participant safety and/or successful completion of the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 0 to 240 minutes after IV methamphetamine
  Blood pressure following IV methamphetamine during treatment with pomaglumetad or placebo
Heart rate | 0 to 240 minutes after IV methamphetamine
  Heart rate following IV methamphetamine during treatment with pomaglumetad or placebo
Rate-pressure product | 0 to 240 minutes after IV methamphetamine
  Rate-pressure product (heart rate * systolic blood pressure, a measure of myocardial oxygen consumption and workload) following IV methamphetamine during treatment with pomaglumetad or placebo
Methamphetamine subjective effects | 0 to 240 minutes after IV methamphetamine
  Self-reported methamphetamine subjective effects assessed with Drug Effect Questionnaire (DEQ-5) and Methamphetamine-based Questionnaire for Stimulant Urges (MA-QSU) following IV methamphetamine during treatment with pomaglumetad or placebo

SECONDARY OUTCOMES:
Peak methamphetamine concentration | 0 to 48 hours after IV methamphetamine
  C-max of methamphetamine during treatment with pomaglumetad or placebo

OTHER OUTCOMES:
Mean choices for methamphetamine | on day of methamphetamine infusion
  Mean choices for methamphetamine during treatment with pomaglumetad or placebo in lab model of methamphetamine self-administration

CONTACTS AND LOCATIONS:
Overall Officials: Keith Heinzerling, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No